CLINICAL TRIAL: NCT00960453
Title: Multiple-dose, Dose Escalation Study to Investigate the Pharmacokinetics/Pharmacodynamics of Sitagliptin in Healthy Male Volunteers
Brief Title: Clinical Trial to Investigate the Pharmacokinetics/Pharmacodynamics of Sitagliptin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Kyung-Sang Yu, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: SNUCPT09_Sitagliptin
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitagliptin 25mg (Other): Repeated administrations for 4 days
  Interventions: Drug: Sitagliptin
- Sitagliptin 50mg (Other): Repeated administrations for 4 days
  Interventions: Drug: Sitagliptin
- Sitagliptin 100mg (Other): Repeated administrations for 4 days
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — Dosage form: 25mg, 50mg ,100mg
  Amount: 25mg, 50mg, 100mg
  Frequency and duration: once a day, for 4 days, including 5 days washout periods

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics and pharmacodynamics of sitagliptin in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 50 years
* A body mass index (BMI) in the range 17-28 kg/m2
* Fasting plasma glucose levels in the range 70-110 mg/dL
* Sufficient ability to understand the nature of the study and any hazards of participating in it
* Provide written informed consent after being fully informed about the study procedures

Exclusion Criteria:

* Presence or history of severe adverse reaction to any drug (e.g., sitagliptin) or a history of severe allergic disease
* Clinically relevant abnormal medical history that could interfere with the objectives of the study
* A subject who has the following screening laboratory test results; creatinine clearance (calculated by Cockcroft-Gault equation) < 80 mL/min
* History of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug
* A subject whose SBP is over 150 mmHg or below 100 mmHg and DBP is over 95 mmHg or below 65 mmHg
* Presence or history of drug abuse
* Participation in other clinical trial within 2 months
* Use of a prescription medicine, herbal medicine within 2 weeks or over-the-counter medication within 1 week before first dose
* Blood donation during 2 months or apheresis during 1 month before the study
* Presence or history of alcohol abuse
* Users of nicotine-containing substances within the previous three months
* Use of grapefruit juice, alcohol or smoking during restriction period
* Subject judged not eligible for study participation by investigator

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics after repeated administrations of sitagliptin 25, 50 and 100 mg | Pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours after drug administration
To evaluate the pharmacodynamics (activity of Dipeptidyl peptidase-IV enzyme) after repeated administrations of sitagliptin 25, 50 and 100 mg | Pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Clinical Trials Center; Seoul National University Hospital, Seoul, South Korea